CLINICAL TRIAL: NCT00013039
Title: Computerized Guidelines Enhanced by Symptoms and History: Clinical Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: CPG 97-001
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Computer reminders

INTERVENTIONS:
Behavioral: Computer reminders

SUMMARY:
Physician compliance with practice guidelines is imperfect. Computer-generated reminders from electronic medical record systems have been shown to increase compliance with guidelines, but they often require symptom and history data, which limits computer facilitation. Heart failure is a serious condition for which compliance with established guidelines is suboptimal. Physicians� compliance with heart failure guidelines may improve if such reminders use symptom and history data.

DETAILED DESCRIPTION:
Background:

Physician compliance with practice guidelines is imperfect. Computer-generated reminders from electronic medical record systems have been shown to increase compliance with guidelines, but they often require symptom and history data, which limits computer facilitation. Heart failure is a serious condition for which compliance with established guidelines is suboptimal. Physicians� compliance with heart failure guidelines may improve if such reminders use symptom and history data.

Objectives:

1) Program standard computer-based guidelines for heart failure using data from the electronic medical record systems at the Indianapolis and Seattle VAMCs. 2) Establish a system for capturing data on symptoms and history from heart failure patients before scheduled primary care visits. 3) Incorporate these data into enhanced computer reminders. 4) Conduct a randomized, controlled trial comparing these two types of reminders� effects on physician prescribing, patient objective and subjective outcomes, and health care utilization.

Methods:

This controlled trial targets patients with objective evidence of left ventricular dysfunction on cardiac imaging studies and a current outpatient diagnosis of heart failure. Primary care physicians in the Indianapolis and Seattle VAMCs have been randomized to receive either standard heart failure treatment reminders or reminders enhanced by history/symptom data. Study data come from the VAMCs electronic medical record systems (i.e., clinical data, utilization, and costs) and patient interviews (heart failure symptoms and medication compliance, heart failure-specific quality of life, and patients� satisfaction with their primary care). Data analysis will be performed at the patient level using general estimating equations to account for patient and physician characteristics and clustering of patients within physicians.

Status:

Data Collection: Enrollment has been completed, with 503 patients enrolled from the Roudebush VAMC in Indianapolis and 250 from the VA Puget Sound Health Care System in Seattle. The trial continues without irregularities in both places. More than 80 percent of eligible patients were enrolled from both sites. Subjective data are being collected prior to scheduled visits on more than 95 percent of enrolled subjects.

ELIGIBILITY:
Inclusion Criteria:

Left ventricular systolic dysfunction by echocardiogram or cardiac MUGA scan and the outpatient diagnosis of heart failure and the primary care physician's statement that he or she is actively treating the patient for heart failure.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Study Completion 2001-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William M. Tierney, MD, Principal Investigator — Richard L. Roudebush VA Medical Center, Indianapolis, IN; Stephan D. Fihn, MD MPH, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (3):
- United States (3):
  - Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

REFERENCES:
- [Result] Subramanian U, Fihn SD, Weinberger M, Plue L, Smith FE, Udris EM, McDonell MB, Eckert GJ, Temkit M, Zhou XH, Chen L, Tierney WM. A controlled trial of including symptom data in computer-based care suggestions for managing patients with chronic heart failure. Am J Med. 2004 Mar 15;116(6):375-84. doi: 10.1016/j.amjmed.2003.11.021. PMID 15006586
- [Result] Udris EM, Au DH, McDonell MB, Chen L, Martin DC, Tierney WM, Fihn SD. Comparing methods to identify general internal medicine clinic patients with chronic heart failure. Am Heart J. 2001 Dec;142(6):1003-9. doi: 10.1067/mhj.2001.119130. PMID 11717604